CLINICAL TRIAL: NCT00525720
Title: Transperineal Interstitial Permanent Brachytherapy Alone for Selected Patients With Intermediate Risk Prostatic Carcinoma
Brief Title: Brachytherapy for Prostatic Carcinoma Patients
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0038; NCI-2012-01594 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-09-04; First posted 2007-09-06 (Estimated); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Prostatic Carcinoma; Intermediate prostate cancer; Transperineal Interstitial Permanent Brachytherapy; Brachytherapy; Prostate brachytherapy; Prostate implant; Prostate; Questionnaire; Survey
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Brachytherapy; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (2):
- Brachytherapy - Participants with < 35% biopsy core (Experimental): Brachytherapy implant procedure lasting 1-2 hours. Questionnaires taking 30 total minutes.
  Interventions: Drug: Brachytherapy; Behavioral: Questionnaire
- Brachytherapy - Participants with > 35% biopsy core (Experimental): Brachytherapy implant procedure lasting 1-2 hours. Questionnaires taking 30 total minutes.
  Interventions: Drug: Brachytherapy; Behavioral: Questionnaire

INTERVENTIONS:
Drug: Brachytherapy — Brachytherapy implant procedure lasting 1-2 hours.
Behavioral: Questionnaire — Questionnaires taking 30 total minutes.
  Other Names: Survey

SUMMARY:
The goal of this clinical research study is to learn if a prostate implant (brachytherapy) can help to control intermediate risk prostate cancer. The safety of this procedure will also be studied.

Prostate brachytherapy is performed by inserting permanent seeds (which are radioactive pellets) into your prostate in order to treat the prostate cancer with radiation therapy.

DETAILED DESCRIPTION:
If you are found to be eligible to take part in this study, you will have an ultrasound of your prostate before brachytherapy so that the prostate can be measured and mapped and the placement of the needles and seeds planned ahead of time. This is a 20-minute outpatient procedure that involves placing a probe (tube) into your rectum, which takes ultrasound pictures of the prostate to learn the size and shape. A specialized radiation plan for each patient is made, and the exact number of needles and seeds depend on the size and shape of the prostate. Ultrasound pictures, using the probe in the rectum, are taken before the implant procedure so that the plan can be made.

Brachytherapy is an outpatient surgical procedure. Under general or spinal anesthesia, you will have thin needles inserted through the skin between the anus and the scrotum. Seeds are inserted into the prostate through the needles. An ultrasound probe (tube which sends images of the prostate to a screen) is placed into the rectum and remains there during the procedure to help direct the needles. After the seeds are inserted, the needles are removed. The seeds remain permanently in the prostate. Typically, about 25 needles are inserted with about 100 seeds. The implant procedure takes about 1-2 hours in the operating room. Afterwards, you will go to the recovery room for 1-3 hours. You will then have a computed tomography (CT) scan after the procedure to make sure the seeds are properly placed. You will then be allowed to return home.

After treatment, you will have a study visit in 4-6 weeks. After that first follow-up visit, you will have follow-up visits at 4, 8, and 12 months (+/- 3 weeks) after treatment. After that, follow-up visits are every 6 months until 5 years after treatment and then once a year from then on (+/- 3 weeks). At these visits, you will have a physical exam. This may include a digital rectal exam if your doctor feels that it is needed. Blood (about 3 teaspoons) will be drawn for routine tests. You will be asked to complete 2 questionnaires about your urinary, bowel, sexual function, and overall quality of life. The 2 questionnaires take about 30 minutes to complete in total. A CT scan of the prostate will also be performed at the first follow-up visit after the implant to make sure the seeds are properly placed.

If blood tests show that your cancer is getting worse, a biopsy may be done after the treatment is complete. A biopsy is done by inserting a needle through the rectum and into the prostate. The procedure is similar to the one done to first diagnose your prostate cancer. Six (6) to 10 samples are usually taken. The doctor will also perform an ultrasound. This is done by placing a tube in the rectum, which shows a picture of the prostate on a screen and is used to guide the biopsies.

You will be taken off study if your disease progresses. Otherwise, you will remain on study indefinitely.

This is an investigational study. Brachytherapy is FDA approved. Up to 300 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of the prostate, clinical stage T1c - T2b (AJCC 6th Edition), N0, M0. Lymph node evaluation by either CT or MRI.
2. Zubrod performance status 0-1.
3. Patient must be greater than or equal to 18 years of age.
4. Patients with intermediate risk prostate cancer as determined by one of the following combinations: Gleason < 7, PSA 10-15; Gleason 7, PSA must be < 10.
5. Prostate specific antigen (PSA) prior to study entry must be less than or equal to 15 ng/ml.
6. Hormone naive.
7. Prostate volumes by TRUS less than or equal to 60 cc.
8. AUA voiding symptom scores </= 15 (alpha blockers allowed); this is completed by the patient.
9. Patients must sign a study-specific informed consent form prior to study entry.

Exclusion Criteria:

1. Stage < T1c, T2c, T3 or T4 disease (AJCC 6th Edition).
2. Lymph node involvement (N1).
3. Evidence of distant metastases (M1).
4. Radical surgery for carcinoma of the prostate, prior pelvic radiation, prior chemotherapy for prostate cancer, prior TURP, prior cryosurgery, TUNA, TUMT of the prostate.
5. Active prostatitis.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2006-08-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Biochemical prostate specific antigen (PSA) progression | 2.5 Years

CONTACTS AND LOCATIONS:
Overall Officials: Steven J. Frank, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org